CLINICAL TRIAL: NCT05427812
Title: A Phase 1/2, First-in-Human, Multicenter, Open-Label, Dose Escalation and Dose-Expansion Study of Single-Agent ISB 1442 in Participants With Relapsed/Refractory Multiple Myeloma
Brief Title: Phase 1/2 Study of ISB 1442 in Relapsed/Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business decision
Sponsor: Ichnos Sciences SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ISB 1442-101
Record Dates: First submitted 2022-06-14; First posted 2022-06-22 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Relapsed/Refractory Multiple Myeloma
Keywords: Open-label; dose-escalation; dose-expansion; ISB 1442; relapsed/refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: Participants will be treated at escalating dose levels in Phase 1 (dose-escalation phase) of the study. Once the safety of ISB 1442 is confirmed and a recommended phase 2 Dose (RP2D) is established in Phase 1, Phase 2 will be initiated for that indication. The Phase 2 design uses the Simon two-stage design with stopping rules for lack of activity, as well as stopping rules for toxicity. Participants will receive ISB 1442, until disease progression, unacceptable toxicity, or any criterion for stopping the study drug or withdrawal from the trial occurs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1: Dose escalation (Experimental): Participants with R/R multiple myeloma (MM) will be administered ISB 1442 weekly by subcutaneous (SC) injection in each 28-day cycle. Dose escalation will begin with an accelerated titration dose escalation and should certain conversion criteria be met, escalation will convert to the standard (3 + 3) dose escalation
  Interventions: Drug: ISB 1442 SC injection escalating doses
- Phase 2 (Dose Expansion): R/R Multiple Myeloma (Experimental): This cohort includes the participants with pathologically confirmed R/R MM and must have received at least 3 prior lines of therapy, including proteasome inhibitors (PIs), immunomodulators (IMiDs), and anti CD38 therapies either in combination or as a single agent; and must not be candidates for regimens known to provide clinical benefit. Participants will receive the recommended Phase 2 Dose (RP2D) of ISB 1442 SC injection determined in Phase 1 of the study for treatment of R/R MM. Each treatment cycle duration is 28 days. The anticipated total duration for each participant will vary, depending on the number of cycles of treatment completed. The treatment phase will extend until participants experience disease progression or unacceptable toxicity, or until any other discontinuation criterion is met.
  Interventions: Drug: ISB 1442 SC injection at RP2D

INTERVENTIONS:
Drug: ISB 1442 SC injection escalating doses — Participants will receive escalating SC doses of ISB 1442
  Arms: Phase 1: Dose escalation
Drug: ISB 1442 SC injection at RP2D — ISB 1442 SC injection dose regimen at RP2D until participants experience disease progression or unacceptable toxicity, or until any other discontinuation criterion is met
  Arms: Phase 2 (Dose Expansion): R/R Multiple Myeloma

SUMMARY:
This study is a first-in-human, Phase 1/2, open label study that will evaluate safety and efficacy of ISB 1442 in relapsed/refractory multiple myeloma (R/R MM).

DETAILED DESCRIPTION:
The study will be conducted in two phases:

* Phase 1: Dose escalation in R/R MM
* Phase 2: Dose expansions in select R/R MM

Participants will be treated at escalating dose levels in Phase 1 (dose-escalation phase) of the study. Once the safety of ISB 1442 is confirmed and a Recommended Phase 2 Dose (RP2D) is established in Phase 1 for a given indication, Phase 2 will be initiated for that indication.

Participants will receive ISB 1442, until disease progression, unacceptable toxicity, or any criterion for stopping the study drug or withdrawal from the trial occurs.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 years or older.
2. Be willing and able to provide written informed consent and any locally required authorization (eg, Health Insurance Portability and Accountability Act of 1996 [HIPAA]) prior to any protocol related procedures, including screening evaluations
3. Phase 1: Patients with pathologically confirmed multiple myeloma (MM) who have progressed on or after standard therapy (relapsed/refractory [R/R] patients):

   1. Must have received at least 3 prior lines of therapy, including PIs, IMiDs, and anti CD38 therapies either in combination or as a single agent; and must not be candidates for regimens known to provide clinical benefit. (Note: Patients in Australia may have received any of the therapies including PIs, IMiDs, and anti CD38 therapies either in combination or as a single agent; and must not be candidates for regimens known to provide clinical benefit ).
   2. Must have measurable M-protein (serum and/or 24-hr urine, or serum free light chains).
4. Phase 2: Patients with pathologically confirmed MM who have progressed on or after standard therapy (R/R patients)
5. Have a body weight ≥ 40.0 kg at screening.
6. Have an Eastern Cooperative Oncology Group (ECOG) performance status score of 2 or less.
7. Have life expectancy of at least 3 months (from date of informed consent signing).
8. Have adequate organ function, including:

   1. Aspartate aminotransferase (AST, GOT) and alanine aminotransferase (ALT, GPT) ≤3.0 × ULN; bilirubin ≤1.5 × ULN. Patients with Gilbert's syndrome may have a bilirubin level >1.5 × ULN, per discussion between the Investigator and medical monitor.
   2. Estimated creatinine clearance ≥45 mL/min as calculated using the Cockcroft-Gault formula or 24-hour urine collection.
9. Left ventricular ejection fraction (LVEF) ≥45% as assessed by echocardiogram (ECHO) or multiple gated acquisition (MUGA) scan.

Exclusion Criteria:

1. Participants with relapsed disease where relapse is characterized only by minimal residual disease parameters (i.e., minimal residual disease positive).
2. Participants with MM with disease where the only measurable parameter is plasmacytoma.
3. Received treatment with anti-CD38 antibodies or CD47 targeted therapies within 1 month of C1D1; systemic anticancer treatments within 14 days before the first dose of study drug (C1D1) or any investigational products within 5 half-lives of C1D1, whichever is appropriate to last therapy received. (eg, non-IMP IMiD, proteasome inhibitor could be considered to be eligible if there is at least 14 days after last dose before C1D1. Note: Treatment with a single course of glucocorticoids is allowed (maximum dose of corticosteroids should not exceed the equivalent of 160 mg [for example, 40 mg/d for 4 days] of dexamethasone). Hormonal therapy for prostate cancer or breast cancer (as adjuvant treatment), and treatment with bisphosphonates and receptor activator of nuclear factor kappa-Β ligand inhibitors are allowed.
4. Received autologous stem cell transplantation within 12 weeks of C1D1.
5. Current participation in another interventional study, including other clinical trials with investigational agents (including investigational vaccines or investigational medical device for disease under study) within 4 weeks of C1D1 and throughout the duration of this trial.
6. Prior radiation therapy within 14 days of C1D1; or prior irradiation to > 25% of the bone marrow. Note: Prophylactic localized ("spot") radiation for areas of pain is allowed.
7. Active malignant central nervous system involvement
8. Known to be refractory to platelet or RBC transfusions
9. Known severe allergic or anaphylactic reactions to human recombinant proteins or excipients used in the ISB 1442 formulation.
10. QTc interval > 480 msec at screening using Fredericia's QT correction formula.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2024-11-19 (Actual)

PRIMARY OUTCOMES:
Phase 1: Frequency and Severity Of Treatment-Emergent Adverse Events (TEAEs) | Up to 18 months
Phase 1: Number of Dose-Limiting Toxicities (DLTS) During the First 28 Days After the First Administration of ISB 1442 (Cycle 1) | Up to 28 days
Phase 2: Multiple Myeloma: Overall Response Rate (ORR) Based on International Myeloma Working Group (IMWG) | 18 months

SECONDARY OUTCOMES:
Maximum Concentration (Cmax) of ISB 1442 in Serum | Up to 28 days
Time to Reach Maximum Concentration (Tmax) of ISB 1442 in Serum | Up to 28 days
Area Under the Concentration Time Curve From Zero to Time t (AUC0-t) of ISB 1442 in Serum | Up to 28 days
Area Under the Concentration Time Curve in Dosing Intervals (AUC0-tau) of ISB1442 in Serum | Up to 28 days
Percent Incidence of Anti-Drug Antibody (ADA) and Neutralizing Antibody (nAb) From Baseline Until End-of-Treatment (EOT) | Baseline to 18 months
Phase 1 and Phase 2: Time to Progression (TTP) | 18 Months
Phase 1 and Phase 2: Time to Next Treatment (TTNT) | 18 Months
Phase 1 and Phase 2: Time to Response (TTR) | 18 Months
Phase 1 and Phase 2: Progression free survival (PFS) | 18 Months
Phase 1 and Phase 2: Overall survival (OS) | 18 Months
Phase 1: Overall Response Rate (ORR) Based on International Myeloma Working Group (IMWG) | 18 months
Phase 1 and Phase 2: Complete Response Rate (CRR) Based on International Myeloma Working Group (IMWG) | 18 months
Phase 1 and Phase 2: Duration of Response (DOR) Based on International Myeloma Working Group (IMWG) | 18 months
Phase 2: Frequency and Severity of Treatment Emergent Adverse Events (TEAEs) | 18 months

CONTACTS AND LOCATIONS:
Locations (15):
- United States (6):
  - University of Miami - Sylvester Comprehensive Cancer Center, Miami, Florida
  - The University of Chicago Medical Center (UCMC) Duchossois Center for Advanced Medicine (DCAM), Chicago, Illinois
  - Barbara Ann Karmanos Cancer Institute - Karmanos Cancer Center - Main Campus, Detroit, Michigan
  - Washington University School of Medicine - Siteman Cancer Center, St Louis, Missouri
  - New York-Presbyterian /Weill Cornell Medical Center - The Myeloma Center, New York, New York
  - Froedtert Hospital & The Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (6):
  - Royal Prince Albert Hospital: Institute of Haematology, Camperdown, New South Wales
  - Pindara Private Hospital, Benowa, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - St. Vincent's Hospital Melbourne, Fitzroy, Victoria
  - The Alfred Hospital-Melbourne, Melbourne, Victoria
  - One Clinical Research Pty Ltd, Nedlands, Western Australia
- India (3):
  - Health Care Global Enterprises Limited (HCG), Bangalore
  - M S Ramaiah Medical College & Hospital, Bangalore
  - Max Super Speciality Hospital, Delhi

IPD SHARING:
Plan to Share IPD: No